CLINICAL TRIAL: NCT01555463
Title: A Randomized, Double-blind, Vehicle-controlled, Multicenter, Parallel-group Clinical Trial to Assess the Safety and Efficacy of Azelaic Acid Foam, 15% Topically Applied Twice Daily for 12 Weeks in Subjects With Papulopustular Rosacea
Brief Title: Safety and Efficacy of Azelaic Acid Foam, 15 % in Papulopustular Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16080; 1401846 (Other: Company Internal)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2023-06-09 (Actual); Status verified 2015-12

CONDITIONS: Papulopustular Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Azelaic acid foam, 15% (BAY39-6251) (Experimental): 0.5 g azelaic acid (AzA) foam, 15% applied twice daily (BID) topical and nonocclusive on facial skin for 12 weeks.
  Interventions: Drug: Azelaic acid foam, 15% (BAY39-6251)
- Vehicle foam (Placebo Comparator): 0.5 g vehicle foam applied twice daily topical and nonocclusive on facial skin for 12 weeks.
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Azelaic acid foam, 15% (BAY39-6251) — Azelaic acid twice daily topical application
  Arms: Azelaic acid foam, 15% (BAY39-6251)
Drug: Vehicle foam — twice daily topical application
  Arms: Vehicle foam

SUMMARY:
The purpose of this study is to assess the safety and efficacy of azelaic acid (AzA) foam, 15% topically applied twice daily for 12 weeks in subjects with papulopustular rosacea compared to its vehicle.

DETAILED DESCRIPTION:
To determine the efficacy of AzA foam, 15% compared to vehicle topically applied twice daily in papulopustular rosacea evaluated by therapeutic success rate according to Investigators Global Assessment (IGA) and change in inflammatory lesion count from baseline to end of treatment.

Evaluation of all adverse events will be covered in Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of papulopustular rosacea
* Free of any clinically significant disease, which could interfere with the study
* Male or female subject aged ≥ 18 years
* Willingness of subject to follow all study procedures
* Signed written informed consent before any study-related activities are carried out

Exclusion Criteria:

* Subjects who are known to be non-responders to azelaic acid
* Presence of dermatoses that might interfere with rosacea diagnosis
* Ocular rosacea; phymatous rosacea; subjects with plaque-type rosacea lesions, papulopustular rosacea that requires systemic treatment
* Topical use of any prescription or non-prescription medication to treat rosacea within 6 weeks prior to randomization and throughout the study
* Systemic use of any prescription or non-prescription medication to treat rosacea (Retinoids within 6 months, Tetracycline within 2 months, Corticosteroids, erythromycin, azithromycin, and/or metronidazole within 4 weeks) prior to randomization and throughout the study
* Facial laser surgery for telangiectasia (or other conditions) within 6 weeks prior to randomization
* Known hypersensitivity to any ingredients of the investigational product formulation
* Participation in another clinical research in parallel or within the last 4 weeks before randomization in this study
* Any condition or therapy that in the investigator's opinion may pose a risk to the subject or that could interfere with any evaluation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 961 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (44):
- United States (44):
  - Birmingham, Alabama
  - Fremont, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Santa Ana, California
  - Santa Monica, California
  - Colorado Springs, Colorado
  - Boynton Beach, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miramar, Florida
  - Ormond Beach, Florida
  - Saint Augustine, Florida
  - Buffalo Grove, Illinois
  - Chicago, Illinois
  - Plainfield, Indiana
  - Louisville, Kentucky
  - Richmond, Kentucky
  - New Orleans, Louisiana
  - Warren, Michigan
  - West Bloomfield, Michigan
  - Fridley, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - East Windsor, New Jersey
  - New York, New York
  - Stony Brook, New York
  - Chapel Hill, North Carolina
  - Hickory, North Carolina
  - High Point, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Johnston, Rhode Island
  - Anderson, South Carolina
  - Knoxville, Tennessee
  - Austin, Texas
  - Plano, Texas
  - Webster, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Spokane, Washington

REFERENCES:
- [Result] Draelos ZD, Elewski BE, Harper JC, Sand M, Staedtler G, Nkulikiyinka R, Shakery K. A phase 3 randomized, double-blind, vehicle-controlled trial of azelaic acid foam 15% in the treatment of papulopustular rosacea. Cutis. 2015 Jul;96(1):54-61. PMID 26244354

RESULTS

PARTICIPANT FLOW:
Period: Treatment
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Started | 483 | 478
Completed | 419 | 399
Not Completed | 64 | 79
Not completed — Adverse Event | 6 | 12
Not completed — Withdrawal by Subject | 24 | 36
Not completed — Lost to Follow-up | 28 | 23
Not completed — Protocol Violation | 4 | 5
Not completed — Other reason | 2 | 3
Period: Follow up
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Started | 447 (Treatment completers and non-completers were asked to participate in the follow-up phase.) | 439 (Treatment completers and non-completers were asked to participate in the follow-up phase.)
Completed | 409 | 394
Not Completed | 38 | 45
Not completed — Adverse Event | 2 | 5
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 22 | 22
Not completed — Lost to Follow-up | 9 | 10
Not completed — Protocol Violation | 2 | 4
Not completed — Other reason | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam | Total
Number analyzed (Participants) | 483 | 478 | 961
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.2 (12.3) | 51.9 (13.2) | 51.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 354 | 348 | 702
  Male | 129 | 130 | 259
Investigator's Global Assessment (IGA) [Number; unit: Participants] — The IGA consists of 5 scores: 1) Clear: no papules and/or pustules; no erythema; 2) Minimal: rare papules and/or pustules; faint up to but not including mild erythema; 3) Mild: few papules and/or pustules; mild erythema; 4) Moderate: pronounced number of papules and/or pustules (but less than numerous papules and/or pustules); moderate erythema; 5) Severe: numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions; moderate to severe erythema.
  Participants
    Clear | 0 | 0 | 0
    Minimal | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 418 | 416 | 834
    Severe | 65 | 62 | 127
Lesion count [Mean (Standard Deviation); unit: Inflammatory lesions] | 21.7 (9.1) | 21.2 (8.7) | 21.4 (8.9)
Erythema rating [Number; unit: Participants]
  Clear or almost clear | 0 | 0 | 0
  Mild | 43 | 39 | 82
  Moderate | 364 | 370 | 734
  Severe | 76 | 69 | 145

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Based Therapeutic Success at End of Treatment (LOCF: Last Observation Carried Forward)
Description: Static evaluation of overall severity of papulopustular rosacea at a given time: 1) Clear: no papules and/or pustules; no erythema; 2) Minimal: rare papules and/or pustules; faint up to but not including mild erythema; 3) Mild: few papules and/or pustules; mild erythema; 4) Moderate: pronounced number of papules and/or pustules (but less than numerous papules and/or pustules); moderate erythema; 5) Severe: numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions; moderate to severe erythema. Therapeutic success is defined as an IGA score of clear or minimal.
Time Frame: At end of treatment (LOCF), up to 12 weeks
Population: All subjects who were randomized and who were dispensed any study medication. For subjects with missing end of treatment observation the last non-missing observation was carried forward, including baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percentage of participants | 32.1 | 23.4
Statistical Analysis 1: Comparison: Azelaic Acid Foam, 15% (BAY39-6251) vs Vehicle Foam; Test type: Superiority or Other; p < .001, Cochran-Mantel-Haenszel; center-adjusted

2. Primary Outcome: Nominal Change From Baseline in Inflammatory Lesion (IL) Count at End of Treatment (LOCF)
Description: The mean (standard deviation) change from baseline in the inflammatory lesion count at the end of treatment is provided.
Time Frame: Baseline and end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Inflammatory lesions | -13.2 (9.5) | -10.3 (9.8)
Statistical Analysis 1: Comparison: Azelaic Acid Foam, 15% (BAY39-6251) vs Vehicle Foam; Test type: Superiority or Other; p < .001, ANCOVA; F-test for treatment effect of the ANCOVA model with treatment group and study center as the factors and baseline lesion count as the covariate

3. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Count at End of Treatment (LOCF)
Description: The mean (standard deviation) percentage change in inflammatory lesion count from baseline to end of study is provided.
Time Frame: Baseline and end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change of inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percent change of inflammatory lesions | -61.6 (33.5) | -50.8 (40.0)

4. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Based Therapeutic Response at End of Treatment (LOCF)
Description: Participants achieving a clear, minimal, or mild IGA at the end of treatment were considered as 'responder'. Participants with an IGA of moderate or severe at the end of treatment were considered as 'non-responder'. Participants who prematurely withdraw from study treatment because of lack of efficacy were coded as 'non-responders'. The percentage of responders is presented.
Time Frame: At end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percentage of participants | 66.3 | 54.4

5. Secondary Outcome: Grouped Changes From Baseline in Erythema Intensity Score at End of Treatment (LOCF)
Description: Erythema was rated as: clear or almost clear; mild; moderate; or severe. For the assessment of the grouped change in erythema ratings, the baseline examination was used to group into 'improved', 'no change', or 'worsened'. A participant was considered to have an 'improved' erythema rating if the erythema rating was lower compared to the baseline rating, 'no change' if the rating was identical, and 'worsened' if the rating was higher. The percentage of participants in each of these categories is presented.
Time Frame: Baseline and end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percentage of participants
  Improved | 61.5 | 51.3
  No change | 36.9 | 46.2
  Worse | 1.7 | 2.5

6. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Scores at End of Treatment (LOCF)
Description: The IGA consists of 5 scores: 1) Clear: no papules and/or pustules; no erythema; 2) Minimal: rare papules and/or pustules; faint up to but not including mild erythema; 3) Mild: few papules and/or pustules; mild erythema; 4) Moderate: pronounced number of papules and/or pustules (but less than numerous papules and/or pustules); moderate erythema; 5) Severe: numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions; moderate to severe erythema. The percentage of participants with each score at the end of treatment is provided.
Time Frame: At end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percentage of participants
  Clear | 4.6 | 4.4
  Minimal | 27.5 | 19.0
  Mild | 34.2 | 31.0
  Moderate | 30.2 | 38.7
  Severe | 3.5 | 6.9

7. Secondary Outcome: Nominal Value of Inflammatory Lesion Count at End of Treatment (LOCF)
Description: The mean (standard deviation) lesion count at the end of treatment is provided.
Time Frame: At end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inflammatory lesions
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Inflammatory lesions | 8.5 (8.9) | 10.8 (11.3)

8. Secondary Outcome: Percentage of Participants With Erythema Intensity Score at End of Treatment (LOCF)
Description: The percentage of participants in each rating category of erythema (clear or almost clear; mild; moderate; severe) at the end of treatment is provided.
Time Frame: At end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percentage of participants
  Clear or almost clear | 9.3 | 8.4
  Mild | 51.8 | 41.8
  Moderate | 34.2 | 43.1
  Severe | 4.8 | 6.7

9. Secondary Outcome: Grouped Changes From Baseline in Telangiectasia Intensity Score at End of Treatment (LOCF)
Description: Telangiectasia was rated as: no; mild; moderate; or severe. At the end of study, a participant was considered to have an 'improved' telangiectasia rating if the telangiectasia rating was lower compared to the baseline rating, 'no change' if the rating was identical, and 'worsened' if the rating was higher. The percentage of participants in each category is presented.
Time Frame: Baseline and end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percentage of participants
  Improved | 27.3 | 22.6
  No change | 65.8 | 69.7
  Worse | 6.8 | 7.7

10. Secondary Outcome: Percentage of Participants With Facial Skin Color Rating at End of Treatment (LOCF)
Description: Facial skin color (as compared with skin outside the treatment area) was rated as: normal; barely visible skin lightening; mild skin lightening; moderate skin lightening; severe skin lightening. The percentage of participants in each category of facial skin color at the end of study is presented.
Time Frame: At end of treatment (LOCF), up to 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 483 | 478
Percentage of participants
  Normal skin color | 80.1 | 78.7
  Barely visible skin-lightening | 8.7 | 10.5
  Mild skin lightening | 8.3 | 7.7
  Moderate skin lightening | 2.7 | 3.1
  Severe skin lightening | 0.2 | 0

11. Secondary Outcome: Participants' Global Assessment of Treatment Response at End of Treatment
Description: At the end of treatment, participants assessed the change of papulopustular rosacea from baseline (how it looked, felt, appeared to others) as excellent improvement, good improvement, fair improvement, no improvement, or worse. The number of participants in each category of this assessment is presented.
Time Frame: At end of treatment, up to 12 weeks
Population: All subjects who were randomized, were dispensed any study medication and had a non-missing observation at end of treatment.
Measure: Number; unit: Participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 432
Participants
  Excellent improvement | 75 | 42
  Good improvement | 174 | 151
  Fair improvement | 121 | 128
  No improvement | 57 | 84
  Worse | 8 | 27

12. Secondary Outcome: Participants' Global Assessment of Tolerability at End of Treatment
Description: At the end of treatment, participants provided their opinion on local tolerability of the investigational product as excellent, good, acceptable despite minor irritation, less acceptable due to continuous irritation, non-acceptable, or no opinion. The number of participants in each category of this assessment is presented.
Time Frame: At end of treatment, up to 12 weeks
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 432
Participants
  Excellent | 167 | 165
  Good | 128 | 173
  Acceptable despite minor irritation | 112 | 49
  Less acceptable due to continuous irritation | 15 | 27
  Not acceptable | 6 | 7
  No opinion | 7 | 11

13. Secondary Outcome: Participants' Opinion on Cosmetic Acceptability at End of Treatment
Description: At the end of treatment, participants provided their opinion on cosmetic acceptability of the investigational product as very good, good, satisfactory, poor, or no opinion. The number of participants in each category of this assessment is presented.
Time Frame: At end of treatment, up to 12 weeks
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 432
Participants
  Very good | 176 | 124
  Good | 112 | 142
  Satisfactory | 95 | 99
  Poor | 36 | 46
  No opinion | 16 | 21

14. Secondary Outcome: Participants' Opinion on Practicability of Product Use in Facial Areas Next to the Hairline at End of Treatment
Description: At the end of treatment, participants provided their opinion on the practicability of the use of the investigational product in facial areas next to the hairline as very good, good, satisfactory, poor, or no opinion. The number of participants in each category of this assessment is presented.
Time Frame: At end of treatment, up to 12 weeks
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 432
Participants
  Very good | 186 | 155
  Good | 143 | 151
  Satisfactory | 67 | 75
  Poor | 14 | 27
  No opinion | 25 | 24

15. Secondary Outcome: Change From Baseline in Rosacea Quality of Life (RosaQoL) Questionnaire at End of Treatment - Overall Quality of Life Score
Description: The Rosacea Quality of Life (RosaQoL) is a questionnaire to evaluate the effect of rosacea on a participant's quality of life. Each of the 21 items in this questionnaire asks about the frequency with which a particular aspect of living with rosacea affects the participant: possible responses for each item are "never" (score=1), "rarely" (score=2), "sometimes" (score=3), "often" (score=4), or "all the time" (score=5). The overall score is the sum of the results from all 21 questions, with possible scores ranging from 21 (best) to 105 (worst); the higher the score, the more quality of life is impaired. The mean (standard deviation) of the change, defined as end of treatment overall score minus baseline overall score, is presented.
Time Frame: Baseline and end of treatment, up to 12 weeks
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 432
Scores on a scale | -6.8 (12.6) | -6.4 (12.1)

16. Secondary Outcome: Number of Participants With Change From Baseline in Dermatology Life Quality Index (DLQI) Questionnaire at End of Treatment - Overall Score
Description: The Dermatology Life Quality Index (DLQI) is a questionnaire consisting of a set of 10 questions that evaluate the degree to which the participant's skin has affected certain behaviors and quality of life over the past week. Possible responses to each question are: "very much" (question 7: "yes") (score=3), "a lot" (score=2), "a little" (score=1), or "not at all"/"not relevant" (score=0). The DLQI overall score is the sum of the results from all 10 questions, with possible scores ranging from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired. The number of participants with score changes (end of treatment - baseline) in DLQI overall score from baseline to end of treatment <=-5 and >-5 are presented.
Time Frame: Baseline and end of treatment, up to 12 weeks
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 431
Participants
  Score change <=-5 | 107 | 82
  Score change >-5 | 328 | 349

17. Secondary Outcome: Change From Baseline in EuroQol Group Questionnaire-Visual Analogue Scale (EQ-VAS) at End of Treatment
Description: The EuroQol Group Questionnaire-Visual Analogue Scale (EQ-VAS) is a standardized instrument for use as a measure of health outcome. The EQ-VAS asks for a judgment of the overall health status assessed by the participant her/himself. The 20-cm visual analog scale (VAS) has endpoints labeled "best imaginable health state" and "worst imaginable health state" that are anchored at 100 and 0, respectively. Respondents are asked to indicate how they rate their own health by drawing a line from an anchor box to that point on the EQ-VAS, which best represents their own health on that day; higher scores indicate a better health state. The median (range) of the change, defined as EQ-VAS at end of treatment minus EQ-VAS at baseline, is presented.
Time Frame: Baseline and end of treatment, up to 12 weeks
Population: as for outcome 11
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 431
Scores on a scale | 0 [-67 to 38] | 0 [-60 to 50]

18. Secondary Outcome: Change From Baseline in Index Value at End of Treatment
Description: The EuroQol Group Questionnaire-5 Dimensions-5 Levels (EQ-5D-5L) is a standardized instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. It is used to assess the level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each dimension is evaluated using 5 levels: "no problems" (level 1), "slight problems" (level 2), "moderate problems" (level 3), "severe problems" (level 4), and "extreme problems" (level 5). A scoring formula developed by EuroQol Group calculates a single index value from the results from all 5 domains along a continuum of 0 (death) to 1 (full health). The median (range) change, defined as the index value at end of treatment minus the index value at baseline, is presented.
Time Frame: Baseline and end of treatment, up to 12 weeks
Population: as for outcome 11
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Number analyzed (Participants) | 435 | 431
Scores on a scale | 0.000 [-0.410 to 0.339] | 0.000 [-0.360 to 0.488]

ADVERSE EVENTS:
Time Frame: From start of treatment until end of study.
Arm/Group | Azelaic Acid Foam, 15% (BAY39-6251) | Vehicle Foam
Serious Adverse Events (participants affected / at risk) | 3/483 | 4/478
Other Adverse Events (participants affected / at risk) | 148/483 | 117/478
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid Foam, 15% (BAY39-6251) (N=483) | Vehicle Foam (N=478)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Accidental death (General disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azelaic Acid Foam, 15% (BAY39-6251) (N=483) | Vehicle Foam (N=478)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 1 (1)
Eyelid bleeding (Eye disorders) | 1 (1) | 0 (0)
Eyelids pruritus (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Application site acne (General disorders) | 0 (0) | 1 (1)
Application site dermatitis (General disorders) | 0 (0) | 2 (2)
Application site dryness (General disorders) | 5 (5) | 3 (3)
Application site erosion (General disorders) | 0 (0) | 1 (4)
Application site erythema (General disorders) | 4 (5) | 4 (4)
Application site exfoliation (General disorders) | 2 (2) | 1 (1)
Application site hypersensitivity (General disorders) | 0 (0) | 1 (1)
Application site inflammation (General disorders) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 3 (4)
Application site pain (General disorders) | 17 (23) | 6 (6)
Application site paraesthesia (General disorders) | 3 (3) | 1 (1)
Application site pruritus (General disorders) | 7 (7) | 2 (2)
Application site reaction (General disorders) | 3 (3) | 0 (0)
Application site scab (General disorders) | 0 (0) | 1 (2)
Application site warmth (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Mycotic allergy (Immune system disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (3) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 2 (3) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (3) | 2 (2)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 3 (3)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (21) | 18 (19)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 3 (3)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 6 (6)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Biopsy lip (Investigations) | 0 (0) | 1 (1)
Biopsy skin (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 21 (25) | 11 (13)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (7)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Morbihan disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Artificial crown procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may publish study results of their own patients only after review/comment by the sponsor. At least 60 days prior to submitting a manuscript to a publisher, a copy of the manuscript will be provided to the sponsor for review. No publication of confidential information shall be made without the sponsor's prior written consent. The PI agrees to delete any confidential information which would prejudice the securing of adequate intellectual property protection from the proposed publication.